CLINICAL TRIAL: NCT01259921
Title: Application of Neurofeedback as a Mechanism of Affect Regulation Treatment of Adults With Complex Adaptation to Chronic Interpersonal Trauma Exposure
Brief Title: EEG Biofeedback in the Treatment of Chronic Treatment-Resistant PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Justice Resource Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ANS2008-06
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2011-06

CONDITIONS: Posttraumatic Stress Disorder
Keywords: EEG biofeedback; neurofeedback; PTSD; Affect Regulation; Chronic Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Neurofeedback

STUDY DESIGN:
Intervention Model Description: EEG Biofeedback versus wait list control condition.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurofeedback T4-P4 (Experimental): 40 sessions of SMR neurofeedback training using T4-P4 placement administered twice weekly
  Interventions: Behavioral: neurofeedback
- Neurofeedback T3-T4 (Active Comparator): 40 sessions of SMR neurofeedback using T3-T4 placement training administered twice weekly
  Interventions: Behavioral: neurofeedback

INTERVENTIONS:
Behavioral: neurofeedback — Operant conditioning of the EEG provided by computer reinforcement.
  Other Names: EEG Spectrum International; Thought Technologies; ProComp 2

SUMMARY:
The purpose of this study is to determine whether neurofeedback (NF) training can significantly reduce the symptoms of Posttraumatic Stress Disorder (PTSD) in individuals with significant affect dysregulation and chronic, treatment-resistant PTSD. The primary aims of this study include:

1. To examine whether NF has the potential to significantly reduce symptoms of PTSD.
2. To examine whether NF training can specifically target the area of affect regulation.
3. To examine the mechanism of NF through elucidating the relationship between affect regulation and PTSD symptom change.

DETAILED DESCRIPTION:
Deficits in affect regulation are associated with a high rate of treatment failure to well-established evidence-based treatments for Posttraumatic Stress Disorder (PTSD), and deficits in this domain are most frequently found in individuals with chronic treatment-resistant PTSD. Aside from one psychological treatment intervention for adult female survivors of child sexual abuse, no published study has targeted improving affect regulation in treatment refractory PTSD. The aim of this study is to test and refine EEG neurofeedback (NF) as an effective treatment for PTSD associated with high levels of affect dysregulation. We believe improved affect regulation will lead to an overall improvement in functioning by addressing deficits in executive functioning in PTSD.

Primary Aim: The primary goal of the research is to refine and evaluate NF training for adults with treatment-resistant PTSD, specifically targeting the domain of affect regulation. We will evaluate the following questions:

1. Will NF decrease chronic PTSD symptoms in a treatment-resistant sample of adults with childhood onset PTSD, as measured with the CAPS and the DTS? Hypothesis 1: Subjects in the active treatment condition will show significantly greater decreases on the CAPS and DTS than subjects in the placebo condition.
2. Will NF improve affect regulation, as measured by the IASC? Hypothesis 2: Subjects in the active treatment condition will show significantly greater improvement on the affect dysregulation subscale of the IASC than individuals in the placebo condition.
3. Will affect regulation, as measured by the IASC, mediate the relationship of NF training and PTSD, as measured with the DTS? Hypothesis 3: The affect dysregulation subscale of the IASC will significantly mediate the relationship between NF and DTS scores while DTS scores will not significantly mediate affect dysregulation.

ELIGIBILITY:
Inclusion Criteria:

* CAPS score of 60 or over
* t-score of 70 or over on the affect dysregulation subscale of the IASC; AND
* Treatment-unresponsiveness as defined by having had at least 3 years of prior treatment focused on dealing with the consequences of the index trauma, or having been in treatment with more than three providers during the preceding decade

Exclusion Criteria:

* Serious non-stable medical illness
* GAF < 40
* Bipolar disorder, obsessive-compulsive disorder (OCD), schizophrenia, and other psychotic disorder, or documented organic impairment
* Active suicidal risk, self-injury or physical aggression toward others within the past year
* Substance dependence or abuse in the past 6 months, as defined by DSM IV criteria
* Individuals taking a benzodiazepine more than twice per week (non-response seen in pilot work) AND
* Any other condition that might interfere with the person's capacity to give informed consent, or to adhere to the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Change in Clinician Administered PTSD Scale Score | Participants are assessed at baseline (prior to beginning training), post-treatment (corresponding to 20 weeks), and at follow-up (1 year post treatment)
  The CAPS is considered the gold standard for the assessment of PTSD (National Center for PTSD Research). It is a clinician administered 30-item interview that corresponds to DSM-IV criteria for PTSD. Each item of the CAPS has two parts, frequency and intensity, which are both scored on a 5-point scale from 0 to 4. A general cut-off rule of frequency greater than or equal to 1 and intensity greater than or equal to 2 for a symptom to count towards diagnosis will be employed in assigning PTSD diagnosis.

SECONDARY OUTCOMES:
Change in Davidson Trauma Scale Score | Participants are assessed at baseline (prior to beginning training), every 4 weeks (corresponding to 8 sessions of training), post-treatment (corresponding to 20 weeks), and at follow-up (1 year post treatment)
  This is a well validated self-report measure of PTSD with clinical reference norms for adults.
Change in Inventory of Altered Self-Capacities Score | Participants are assessed at baseline (prior to beginning training), every 4 weeks (corresponding to 8 sessions of training), post-treatment (corresponding to 20 weeks), and at follow-up (1 year post treatment)
  The IASC is a 63-item standardized measure of disturbed functioning in relation to self and others. The IASC measures seven domains of functioning: Interpersonal Conflicts, Idealization-Disillusionment, Abandonment Concerns, Identity Impairment, Susceptibility to Influence, Affect Dysregulation, and Tension Reduction Activities.

CONTACTS AND LOCATIONS:
Overall Officials: Bessel van der Kolk, M.D., Principal Investigator — Justice Resource Institute; Mark Gapen, Ph.D., Study Director — Justice Resource Institute
Locations (1):
- the Trauma Center at JRI, Brookline, Massachusetts, United States

REFERENCES:
- [Background] Gapen M, van der Kolk BA, Hamlin E, Hirshberg L, Suvak M, Spinazzola J. A Pilot Study of Neurofeedback for Chronic PTSD. Appl Psychophysiol Biofeedback. 2016 Sep;41(3):251-61. doi: 10.1007/s10484-015-9326-5. PMID 26782083